CLINICAL TRIAL: NCT01787929
Title: Cemented Versus Uncemented Hemiarthroplasty for Displaced Femoral Neck Fracture in Elderly Patient : a Randomized Prospective Trial
Brief Title: Displaced Femoral Neck Fracture in Elderly Patient. Should Cement be Used for Hip Hemiarthroplasty ?
Acronym: PIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 12-PP-10
Record Dates: First submitted 2013-01-17; First posted 2013-02-11 (Estimated); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Hemiarthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cemented hemiarthroplasty (Other): hemiarthroplasty surgery with cement for displaced femoral neck fractures
  Interventions: Procedure: hemiarthroplasty for displaced femoral neck fractures
- Uncemented hemiarthroplasty (Other): hemiarthroplasty surgery without cement is a surgery for displaced femoral neck fractures
  Interventions: Procedure: hemiarthroplasty for displaced femoral neck fractures

INTERVENTIONS:
Procedure: hemiarthroplasty for displaced femoral neck fractures — Hemiarthroplasty is a surgery for displaced femoral neck fractures

SUMMARY:
The purpose of this study was to identify the clinical relevance of cementless hemiarthroplasties, compare Harris functional score.The hypothesis is the non-inferiority of cementless hemiarthroplasties compare cemented hemiarthroplasties in order to justify the relevance of cementless hemiarthroplasties in displaced femoral neck fractures.

150 patients will be included, 75 with cemented hemiarthroplasty and 75 with uncemented hemiarthroplasty. They will be followed during one year after the surgery, with a functionality assessment at 3 month and 12 month.

DETAILED DESCRIPTION:
Most subcapital femoral neck fractures occur in the elderly population and are the result of low-energy trauma. Return of the patient to prefracture level of function usually can best be accomplished with surgery. Nonsurgical management has resulted in an excessive rate of medical morbidity and mortality. The overall 1-year mortality rate after hip fracture in the elderly ranges from 14% to 36%.

Prosthetic replacement has been favored for the treatment of displaced femoral neck fractures in the frail, elderly population with multiple medical comorbidities because of the challenges of achieving stable proximal fragment fixation in osteopenic bone, and the need for early, full weight-bearing mobilization. Failure rates of 30% to 40% have been consistently reported over multiple series over the past few decades in elderly patients with displaced femoral neck fractures treated with internal fixation.

Once prosthetic arthroplasty has been chosen, further controversy surrounds the type of fixation, cemented or cementless. Good to excellent results can be expected with either cemented or cementless newer generation arthroplasties. Risks of cementless arthroplasty include femoral fracture, prosthesis subsidence, and anterior thigh pain. Cementation of the prosthesis places the patient at risk for intraoperative death or embolization of marrow content during cementation.

The aim of the study is to assess the clinical relevance of a collared uncemented stem compared with use of cemented stem in elderly population with displaced femoral neck fracture.

A randomised trial will include 150 patients with an acute displaced femoral neck fracture in an elderly population. All patient will give informed consent, and the research protocol is approved by the regional ethics committee. The inclusion criteria are an age of at least 70 years old, a displaced femoral neck fracture (Garden stage III or IV), an ASA grade< 4, ambulatory and non cognive impairment patients. Clinical and radiographic examinations will be perform at perioperative period, at 3 and 12 month after surgery. The main outcome measures will be functional score, pain, mobility, complications, reoperations, activity of daily living, quality of life, strenght, and radiolographic subsidence.

The primary hypothesis of this study is that use of a collared uncemented stem would not provide an improvement in functional outcome compared with use of cemented stem in elderly population with displaced femoral neck fracture.

ELIGIBILITY:
Inclusion Criteria:

* displaced femoral neck fractures (Garden III and IV)
* 70 year old or more
* ASA score < or = III
* Lee score < or = 2

Exclusion Criteria:

* Parker score <4
* pathological femoral neck fracture ( paget disease or tumor)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 170 (Actual)
Dates: Start 2016-02-07 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Functionality | Changes at 3 and 12 month post-operative
  Functionality will be assessed at 3 and 12 month after surgery by Harris test scoring.

CONTACTS AND LOCATIONS:
Overall Officials: Regis BERNARD DE DOMPSURE, MD, Principal Investigator — University Nice Hospital
Locations (1):
- orthopedics department, University Hospital, Nice, France